CLINICAL TRIAL: NCT01607112
Title: A Phase III Study for Evaluation of Immunogenicity and Reactogenicity of Fluarix/Influsplit SSW 2012/2013 in People Aged 18 Years and Above
Brief Title: A Study for Evaluation of Immunogenicity and Reactogenicity of Fluarix/Influsplit SSW 2012/2013 in People Aged 18 Years and Above
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 116663; 2012-000789-39 (EudraCT Number)
Record Dates: First submitted 2012-05-24; First posted 2012-05-28 (Estimated); Results first posted 2013-12-06 (Estimated); Last update posted 2018-09-07 (Actual); Status verified 2013-11

CONDITIONS: Influenza
Keywords: Influenza; Healthy; Immunogenicity; Elderly; Safety; Adults
MeSH Terms: conditions — Influenza, Human | interventions — fluarix

ARMS (2):
- Fluarix/Influsplit 18-60 Years Group (Experimental): Subjects 18-60 years of age received 1 dose of Fluarix/Influsplit SSW 2012-2013 vaccine at Day 0. The vaccine was administered intramuscularly in the deltoid of the non-dominant arm.
  Interventions: Biological: Fluarix/Influsplit SSW 2012-2013
- Fluarix/Influsplit > 60 Years Group (Experimental): Subjects above 60 years of age received 1 dose of Fluarix/Influsplit SSW 2012-2013 vaccine at Day 0. The vaccine was administered intramuscularly in the deltoid of the non-dominant arm.
  Interventions: Biological: Fluarix/Influsplit SSW 2012-2013

INTERVENTIONS:
Biological: Fluarix/Influsplit SSW 2012-2013 — 1 dose administered intramuscularly (or deeply subcutaneously) in the deltoid region of the non-dominant arm

SUMMARY:
The purpose of this study is to assess the immunogenicity and safety of GSK Biologicals' trivalent influenza vaccine manufactured for the 2012/2013 influenza season administered in adults (18 to 60 years) and in elderly (over 60 years).

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes can and will comply with the requirements of the protocol.
* A male or female aged 18 years or above at the time of vaccination.
* Written informed consent obtained from the subject.
* Healthy subjects or subjects with well-controlled chronic diseases as established by medical history and clinical examination before entering the study.
* Female subjects of non-childbearing potential may be enrolled in the study.
* Female subjects of childbearing potential may be enrolled in the study, if the subject:

  * has practiced adequate contraception for 30 days prior to vaccination, and
  * has a negative pregnancy test on the day of vaccination, and
  * has agreed to continue adequate contraception during the entire treatment period and for 2 months after completion of vaccination.

Exclusion Criteria:

* Use of any investigational or non-registered product other than the study vaccine within 30 days preceding the dose of study vaccine, or planned use during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs within the six months prior to vaccination. Inhaled and topical steroids are allowed.
* Administration of immunoglobulins and/or any blood products within the three months preceding the administration of the study vaccine or planned administration during the study period.
* Administration of an influenza vaccine within the six months preceding the study vaccination.
* Planned administration/ administration of a vaccine other than the study vaccine within 30 days before study vaccination and during the entire study period.
* Clinically or virologically confirmed influenza infection within the six months preceding the study vaccination.
* Acute disease and/or fever at the time of enrolment.
* Acute, clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination or laboratory screening tests.
* Chronic underlying disease, not stabilized or clinically serious.
* History of chronic alcohol consumption and/or drug abuse.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* History of Guillain-Barré syndrome.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* Anaphylaxis following the administration of vaccine(s).
* Pregnant or lactating female.
* Female planning to become pregnant or planning to discontinue contraceptive precautions.
* Any condition which, in the opinion of the investigator, prevents the subject from participating in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2012-07-10; Primary Completion 2012-07-31 (Actual); Study Completion 2012-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Dresden, Saxony, Germany

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Approximately 50% of subjects in the Fluarix/Influsplit > 60 Years Group and a maximum of 25% of subjects in the Fluarix/Influsplit 18-60 Years Group were allowed to have had a seasonal influenza vaccination the year before.
Period: Overall Study
Arm/Group | Fluarix/Influsplit 18-60 Years Group | Fluarix/Influsplit > 60 Years Group
Started | 60 | 59
Completed | 60 | 59
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fluarix/Influsplit 18-60 Years Group | Fluarix/Influsplit > 60 Years Group | Total
Number analyzed (Participants) | 60 | 59 | 119
Age, Continuous [Mean (Standard Deviation); unit: Years] | 35.7 (11.98) | 70.3 (5.87) | 52.8 (19.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 34 | 64
  Male | 30 | 25 | 55

OUTCOME MEASURES:

1. Primary Outcome: Humoral Immune Response in Terms of Haemagglutination (HA) Antibody Titers Against Each of the Three Vaccine Influenza Strains
Description: Antibody titers were expressed as Geometric mean titers (GMTs). The vaccine strains assessed were Flu A/Christchurch/16/10 (H1N1), Flu A/Victoria/361/11 (H3N2) and Flu B/Hubei-Wujiagang/158/09 (Yamagata).
Time Frame: At Day 0 and Day 21
Population: Analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity which included all evaluable subjects for whom data concerning immunogenicity outcome measures were available.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Fluarix/Influsplit 18-60 Years Group | Fluarix/Influsplit > 60 Years Group
Number analyzed (Participants) | 59 | 58
Titer
  H1N1, Day 0 | 20.57 [13.98 to 30.27] | 19.02 [14.35 to 25.22]
  H1N1, Day 21 | 366.04 [264.22 to 507.09] | 110.44 [79.50 to 153.43]
  H3N2, Day 0 | 16.17 [12.07 to 21.65] | 23.90 [17.07 to 33.45]
  H3N2, Day 21 | 93.19 [73.75 to 117.76] | 65.63 [48.37 to 89.05]
  Yamagata, Day 0 | 68.60 [50.26 to 93.63] | 70.19 [58.98 to 83.53]
  Yamagata, Day 21 | 431.85 [332.61 to 560.70] | 223.56 [183.62 to 272.19]

2. Primary Outcome: Number of Subjects Who Were Seroprotected for Anti-HA Antibodies Against Each of the Three Vaccine Influenza Strains.
Description: Seroprotection rate (SPR) was defined as the number of vaccinees with serum haemagglutination inhibition (HI) titer greater than or equal to (≥) 1:40.
Time Frame: At Day 0 and Day 21
Population: as for outcome 1
Measure: Number; unit: Subjects
Groups:
- Fluarix/Influsplit 18-60 Years Group: Subjects 18-60 years of age received 1 dose of Fluarix/Influsplit SSW 2012-2013 at Day 0. The vaccine was administered intramuscularly in the deltoid of the non-dominant arm.
- Fluarix/Influsplit > 60 Years Group: Subjects above 60 years of age received 1 dose of Fluarix/Influsplit SSW 2012-2013 at Day 0. The vaccine was administered intramuscularly in the deltoid of the non-dominant arm.
Arm/Group | Fluarix/Influsplit 18-60 Years Group | Fluarix/Influsplit > 60 Years Group
Number analyzed (Participants) | 59 | 58
Subjects
  H1N1, Day 0 | 20 | 14
  H1N1, Day 21 | 55 | 47
  H3N2, Day 0 | 15 | 23
  H3N2, Day 21 | 51 | 41
  Yamagata, Day 0 | 42 | 51
  Yamagata, Day 21 | 59 | 58

3. Primary Outcome: Number of Seroconverted Subjects for Anti-HA Antibodies Against Each of the Three Vaccine Influenza Strains.
Description: A seroconverted subjects was defined as a vaccinee with either a pre-vaccination titer less than (<) 1:10 and a post-vaccination titer ≥ 1:40, or a pre-vaccination titer ≥ 1:10 and at least a 4-fold increase in post-vaccination titer.
Time Frame: At Day 21
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Fluarix/Influsplit 18-60 Years Group | Fluarix/Influsplit > 60 Years Group
Number analyzed (Participants) | 59 | 58
Subjects
  H1N1 | 45 | 34
  H3N2 | 34 | 14
  Yamagata | 38 | 24

4. Primary Outcome: Mean Geometric Increase (MGI) for Haemagglutination Inhibition (HI) Antibody Titer Against Each of the Three Vaccine Influenza Strains.
Description: MGI was defined as the fold increase in serum HI GMT post-vaccination compared to Day 0.
Time Frame: At Day 21
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Fold increase
Arm/Group | Fluarix/Influsplit 18-60 Years Group | Fluarix/Influsplit > 60 Years Group
Number analyzed (Participants) | 59 | 58
Fold increase
  H1N1 | 17.8 [11.5 to 27.6] | 5.8 [4.2 to 8.0]
  H3N2 | 5.8 [4.2 to 7.8] | 2.7 [2.2 to 3.4]
  Yamagata | 6.3 [4.6 to 8.7] | 3.2 [2.6 to 3.9]

5. Primary Outcome: Number of Subjects With Seroprotection Power (SPP) for HI Antibody Titer Against Each of the Three Vaccine Influenza Strains Above the Cut-off Value.
Description: SPP was defined as the number of vaccinees with a pre-vaccination titer < 1:40 and a post-vaccination titer ≥ 1:40.
Time Frame: At Day 21
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Fluarix/Influsplit 18-60 Years Group | Fluarix/Influsplit > 60 Years Group
Number analyzed (Participants) | 44 | 44
Subjects
  H1N1 [N=39,44] | 35 | 33
  H3N2 [N=44,35] | 36 | 18
  Yamagata [N=17,7] | 17 | 7

6. Secondary Outcome: Humoral Immune Response in Terms of Anti-HA Antibodies Against Each of the Three Vaccine Influenza Strains.
Description: Antibody titers were expressed as Geometric mean titers (GMTs). The vaccine strains included H1N1, H3N2 and Yamagata antigens. The outcome measure was assessed by influenza vaccination status in the 2011-2012 season, in subjects aged greater than (>) 60 years.
Time Frame: At Day 0 and Day 21
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Groups:
- Fluarix/Influsplit > 60 Years Group With Vaccination: Subjects above 60 years of age received 1 dose of Fluarix/Influsplit SSW 2012-2013 vaccine at Day 0 and who had received seasonal Flu vaccination in 2011-2012. The vaccine was administered intramuscularly in the deltoid of the non-dominant arm.
- Fluarix/Influsplit > 60 Years Group Without Vaccination: Subjects above 60 years of age received 1 dose of Fluarix/Influsplit SSW 2012-2013 vaccine at Day 0 and did not receive seasonal Flu vaccination in 2011-2012. The vaccine was administered intramuscularly in the deltoid of the non-dominant arm.
Arm/Group | Fluarix/Influsplit > 60 Years Group With Vaccination | Fluarix/Influsplit > 60 Years Group Without Vaccination
Number analyzed (Participants) | 30 | 28
Titer
  H1N1, Day 0 | 22.13 [14.86 to 32.95] | 16.18 [10.67 to 24.53]
  H1N1, Day 21 | 92.92 [59.75 to 144.52] | 132.89 [79.80 to 221.30]
  H3N2, Day 0 | 24.02 [15.11 to 38.17] | 23.76 [14.12 to 40.00]
  H3N2, Day 21 | 57.22 [35.97 to 91.03] | 76.01 [50.24 to 114.99]
  Yamagata, Day 0 | 77.34 [62.16 to 96.23] | 63.26 [47.63 to 84.01]
  Yamagata, Day 21 | 208.70 [159.83 to 272.52] | 240.65 [177.18 to 326.87]

7. Secondary Outcome: Number of Subjects Who Were Seroprotected for Anti-HA Antibodies Against Each of the Three Vaccine Influenza Strains.
Description: Seroprotection rate SPR was defined as the number of vaccinees with serum haemagglutination inhibition (HI) titer greater than or equal to (≥) 1:40. The outcome measure was assessed by the influenza vaccination status in the 2011-2012 season, in subjects aged > 60 years.
Time Frame: At Day 0 and Day 21
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Fluarix/Influsplit > 60 Years Group With Vaccination | Fluarix/Influsplit > 60 Years Group Without Vaccination
Number analyzed (Participants) | 30 | 28
Subjects
  H1N1, Day 0 | 9 | 5
  H1N1, Day 21 | 24 | 23
  H3N2, Day 0 | 12 | 11
  H3N2, Day 21 | 21 | 20
  Yamagata, Day 0 | 28 | 23
  Yamagata, Day 21 | 30 | 28

8. Secondary Outcome: Number of Subjects Who Seroconverted for Anti-HA Antibodies Against Each of the Three Vaccine Influenza Strains.
Description: SCR was defined as the number of vaccinees with either a pre-vaccination titer less than (<) 1:10 and a post-vaccination titer ≥ 1:40, or a pre-vaccination titer ≥ 1:10 and at least 4-fold increase in post-vaccination titer. The outcome measure was assessed by influenza vaccination status in the 2011-2012 season, in subjects aged > 60 years.
Time Frame: At Day 21
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Fluarix/Influsplit > 60 Years Group With Vaccination | Fluarix/Influsplit > 60 Years Group Without Vaccination
Number analyzed (Participants) | 30 | 28
Subjects
  H1N1 | 15 | 19
  H3N2 | 6 | 8
  Yamagata | 11 | 13

9. Secondary Outcome: Mean Geometric Increase (MGI) for Haemagglutination Inhibition (HI) Antibody Titer Against Each of the Three Vaccine Influenza Strains.
Description: MGI was defined as the fold increase in serum HI GMT post-vaccination compared to Day 0. This outcome measure was assessed by influenza vaccination status in the 2011-2012 season, in subjects aged > 60 years.
Time Frame: At Day 21
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Fold increase
Arm/Group | Fluarix/Influsplit > 60 Years Group With Vaccination | Fluarix/Influsplit > 60 Years Group Without Vaccination
Number analyzed (Participants) | 30 | 28
Fold increase
  H1N1 | 4.2 [2.8 to 6.4] | 8.2 [5.1 to 13.3]
  H3N2 | 2.4 [1.9 to 3.0] | 3.2 [2.1 to 4.8]
  Yamagata | 2.7 [2.2 to 3.4] | 3.8 [2.8 to 5.3]

10. Secondary Outcome: Duration of Solicited Local Symptoms.
Description: Duration was defined as number of days with any grade of local symptoms.
Time Frame: During the 4-day follow-up period (Days 0-3) after vaccination
Population: Analysis was performed on the Total Vaccinated cohort, which included all subjects with vaccine administration documented.
Measure: Median (Full Range); unit: Days
Arm/Group | Fluarix/Influsplit 18-60 Years Group | Fluarix/Influsplit > 60 Years Group
Number analyzed (Participants) | 33 | 23
Days
  Induration [N=2,4] | 2.5 [2.0 to 3.0] | 2.0 [1.0 to 2.0]
  Pain [N=33,23] | 2.0 [1.0 to 4.0] | 2.0 [1.0 to 3.0]
  Redness [N=6,7] | 2.5 [1.0 to 4.0] | 2.0 [1.0 to 3.0]
  Swelling [N=6,5] | 2.0 [1.0 to 4.0] | 2.0 [1.0 to 3.0]

11. Secondary Outcome: Number of Subjects Reporting Any and Grade 3 Solicited Local Symptoms.
Description: Solicited local symptoms assessed were ecchymosis, induration, pain, redness and swelling. Any was defined as any solicited local symptom reported irrespective of intensity. Grade 3 pain was defined as pain that prevented normal everyday activities. Grade 3 ecchymosis, induration, redness and swelling was greater than 100 millimeters (mm) i.e. >100mm.
Time Frame: During the 4-day (Day 0-Day 3) follow-up period after vaccination
Population: Analysis was performed on the Total Vaccinated cohort which included all subjects with vaccine administration documented.
Measure: Number; unit: Subjects
Arm/Group | Fluarix/Influsplit 18-60 Years Group | Fluarix/Influsplit > 60 Years Group
Number analyzed (Participants) | 60 | 59
Subjects
  Any Ecchymosis | 0 | 0
  Grade 3 Ecchymosis | 0 | 0
  Any Induration | 2 | 4
  Grade 3 Induration | 0 | 0
  Any Pain | 33 | 23
  Grade 3 Pain | 1 | 0
  Any Redness | 6 | 7
  Grade 3 Redness | 0 | 0
  Any Swelling | 6 | 5
  Grade 3 Swelling | 0 | 0

12. Secondary Outcome: Duration of Solicited General Symptoms.
Description: Duration was defined as number of days with any grade of general symptoms.
Time Frame: During the 4-day follow-up period (Days 0-3) after vaccination
Population: as for outcome 10
Measure: Median (Full Range); unit: Days
Arm/Group | Fluarix/Influsplit 18-60 Years Group | Fluarix/Influsplit > 60 Years Group
Number analyzed (Participants) | 15 | 14
Days
  Arthralgia [N=2,4] | 2.5 [2.0 to 3.0] | 3.0 [1.0 to 4.0]
  Fatigue [N=11,14] | 1.0 [1.0 to 3.0] | 2.0 [1.0 to 4.0]
  Gastrointestinal symptoms [N=4,3] | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 2.0]
  Headache [N=15,7] | 1.0 [1.0 to 4.0] | 1.0 [1.0 to 1.0]
  Myalgia [N=11,7] | 1.0 [1.0 to 3.0] | 1.0 [1.0 to 4.0]
  Sweating increase [N=8,9] | 1.0 [1.0 to 4.0] | 2.0 [1.0 to 4.0]
  Shivering [N=1,2] | 1.0 [1.0 to 1.0] | 1.5 [1.0 to 2.0]
  Fever (Axillary) [N=2,1] | 1.0 [1.0 to 1.0] | 4.0 [4.0 to 4.0]

13. Secondary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Solicited General Symptoms.
Description: Solicited general symptoms assessed were arthralgia, fatigue, gastrointestinal symptoms, headache, myalgia, shivering, increased sweating and fever [axillary temperature above 37.5 degrees Celsius (°C)]. Gastrointestinal symptoms included nausea, vomiting, diarrhea and/or abdominal pain.
  Any = any solicited general symptom reported irrespective of intensity and relationship to vaccination. Related = symptoms considered by the investigator to have a causal relationship to vaccination. Grade 3 symptoms = symptoms that prevented normal activity. Grade 3 fever = axillary temperature above 39.0°C
Time Frame: During the 4-day follow-up period (Day 0-3) after vaccination
Population: as for outcome 10
Measure: Number; unit: Subjects
Arm/Group | Fluarix/Influsplit 18-60 Years Group | Fluarix/Influsplit > 60 Years Group
Number analyzed (Participants) | 60 | 59
Subjects
  Any Arthralgia | 2 | 4
  Grade 3 Arthralgia | 0 | 0
  Related Arthralgia | 2 | 1
  Any Fatigue | 11 | 14
  Grade 3 Fatigue | 1 | 0
  Related Fatigue | 7 | 10
  Any Gastrointestinal symptoms | 4 | 3
  Grade 3 Gastrointestinal symptoms | 0 | 0
  Related Gastrointestinal symptoms | 2 | 3
  Any Headache | 15 | 7
  Grade 3 Headache | 1 | 1
  Related Headache | 11 | 6
  Any Myalgia | 11 | 7
  Grade 3 Myalgia | 0 | 0
  Related Myalgia | 11 | 5
  Any Shivering | 1 | 2
  Grade 3 Shivering | 0 | 0
  Related Shivering | 1 | 1
  Any Sweating increase | 8 | 9
  Grade 3 Sweating increase | 0 | 0
  Related Sweating increase | 6 | 6
  Any Fever ≥37.5°C | 2 | 1
  Grade 3 Fever >39.0°C | 0 | 0
  Related Fever | 2 | 1

14. Secondary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Unsolicited Adverse Events (AEs).
Description: Unsolicited AE covers any AE reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as occurrence of any unsolicited symptom regardless of intensity grade or relation to vaccination. Grade 3 was an event that prevented normal activities and related was defined as an unsolicited AE assessed by the investigator to be causally related to the study vaccination.
Time Frame: During the 21-day follow-up period (Days 0-20) after vaccination
Population: as for outcome 10
Measure: Number; unit: Subjects
Arm/Group | Fluarix/Influsplit 18-60 Years Group | Fluarix/Influsplit > 60 Years Group
Number analyzed (Participants) | 60 | 59
Subjects
  Any Unsolicted AEs | 8 | 11
  Grade 3 Unsolicted AEs | 0 | 1
  Related Unsolicted AEs | 4 | 3

15. Secondary Outcome: Number of Subjects Reporting Any and Related Serious Adverse Events (SAEs)
Description: A serious adverse event was any untoward medical occurrence that: resulted in death, was life-threatening, required hospitalization or prolongation of existing hospitalization, resulted in disability/incapacity or was a congenital anomaly/birth defect in the offspring of a study subject. Any was defined as occurrence of any symptom regardless of intensity grade or relation to vaccination and related was an event assessed by the investigator as causally related to the study vaccination.
Time Frame: During the entire study period (Days 0-21)
Population: as for outcome 10
Measure: Number; unit: Subjects
Arm/Group | Fluarix/Influsplit 18-60 Years Group | Fluarix/Influsplit > 60 Years Group
Number analyzed (Participants) | 60 | 59
Subjects
  Any SAEs | 0 | 0
  Related SAEs | 0 | 0

ADVERSE EVENTS:
Time Frame: Serious Adverse Events: From Day 0 to Day 21; Solicited local and general symptoms: During the 4-day (Days 0-3) post-vaccination period; Unsolicited symptoms: During the 21-day (Day 0-20) post-vaccination period
Groups:
- Adult Group: Subjects 18-60 years of age received 1 dose of Fluarix/Influsplit SSW 2012-2013 vaccine at Day 0. The vaccine was administered intramuscularly in the deltoid of the non-dominant arm.
- Elderly Group: Subjects above 60 years of age received 1 dose of Fluarix/Influsplit SSW 2012-2013 vaccine at Day 0. The vaccine was administered intramuscularly in the deltoid of the non-dominant arm.
Arm/Group | Adult Group | Elderly Group
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/59
Other Adverse Events (participants affected / at risk) | 39/60 | 35/59
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Adult Group (N=60) | Elderly Group (N=59)
Induration (General disorders) | 2 | 4
Pain (General disorders) | 33 | 23
Redness (General disorders) | 6 | 7
Swelling (General disorders) | 6 | 5
Arthralgia (General disorders) | 2 | 4
Fatigue (General disorders) | 11 | 14
Gastrointestinal symptoms (General disorders) | 4 | 3
Headache (General disorders) | 15 | 7
Myalgia (General disorders) | 11 | 7
Sweating increase (General disorders) | 8 | 9
Injection site pruritus (General disorders) | 3 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.